CLINICAL TRIAL: NCT05727527
Title: The Effect of Using a Sugar-free Candy Flavoring Before Local Anesthesia Injection on Anxiety and Pain Perception in Children: a Split-mouth Randomized Clinical Trial
Brief Title: Effect of a Candy Flavoring Before Local Anesthesia on Anxiety and Pain Perception in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 692l2021
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Local Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Will initially receive the infiltration injection after applying a candy flavor first, followed by sterile water in the next visit
  Interventions: Procedure: Local Anesthesia 1; Procedure: Local Anesthesia 2
- Control group (Active Comparator): Will initially receive the infiltration injection after applying sterile water first, followed by candy flavor in the next visit
  Interventions: Procedure: Local Anesthesia 1; Procedure: Local Anesthesia 2

INTERVENTIONS:
Procedure: Local Anesthesia 1 — Local anesthesia injection after applying a candy flavor
Procedure: Local Anesthesia 2 — Local anesthesia injection after applying sterile water

SUMMARY:
This is a randomized clinical trial that aimed to test the effect of using sugar-free flavors as a sensory distraction technique during local anesthesia on pain perception when compared to a negative control group. Applying the flavor before injecting local anesthesia helped in distracting the child and reduced the associated pain.

DETAILED DESCRIPTION:
Background: Distraction techniques can be very useful in managing children on the dental chair and to guide their attention away from a painful stimulus. No studies so far have used a sugar-free solution as a distraction method.

Aim: To test the effect of using sugar-free flavors as a sensory distraction technique during local anesthesia on pain perception and anxiety when compared to negative control group, using a split-mouth randomized study design.

Methods: A total of 84 children, aged 4-9 years with no previous dental experience and require the same treatment on the upper primary first or second molars bilaterally were included in this study. Each child received two injections. The children were randomly allocated into two groups, group 1 received the first injection after applying a flavor, and group 2 received the first injection after applying sterile water. The children received the first injection either on the right or left side, and switched sides on the next visit, resulting in (n=168) total injections. The observed pain perception was assessed using the SEM scale. Wong-Baker Faces pain rating scale will be used to assess the pain reported by the child. Pulse rate, BMI, and sweet taste preference were also recorded by an independent observer to ensure blinding.

Results: Using a sugar-free candy flavor before injecting local anesthesia helps in reducing pain accompanying local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (ASA Grade 1 status) children
* First dental experience for the child including local anesthesia.
* Children with caries lesions that require restorative treatment.
* Children who require the same treatment on upper primary first or second molars bilaterally.

Exclusion Criteria:

* Children with poor behavior (unable to cooperate for dental treatment).
* Previous unpleasant dental experience (dental phobia).
* History of abscess, redness, fistula in the injection site (need for extraction).
* Presence of a systemic disease, mental, cognitive and intellectual disabilities.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Pain score | During injection
  Reported pain by the child will be assessed using the Wong-Baker Faces Pain Rating Scale, Scores range from 0-10, higher scores mean more pain

SECONDARY OUTCOMES:
Anxiety | Before and during injection
  Anxiety will be assessed through pulse rate measurements recorded before, during and the injection using a fingertip pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Ola B. Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Ola B. Al-Batayneh, Irbid, Jordan

REFERENCES:
- [Background] Alanazi KJ, Pani S, AlGhanim N. Efficacy of external cold and a vibrating device in reducing discomfort of dental injections in children: A split mouth randomised crossover study. Eur Arch Paediatr Dent. 2019 Apr;20(2):79-84. doi: 10.1007/s40368-018-0399-8. Epub 2018 Dec 5. PMID 30519955
- [Background] Al-Khotani A, Bello LA, Christidis N. Effects of audiovisual distraction on children's behaviour during dental treatment: a randomized controlled clinical trial. Acta Odontol Scand. 2016 Aug;74(6):494-501. doi: 10.1080/00016357.2016.1206211. Epub 2016 Jul 13. PMID 27409593
- [Background] Asvanund Y, Mitrakul K, Juhong RO, Arunakul M. Effect of audiovisual eyeglasses during local anesthesia injections in 5- to 8-year-old children. Quintessence Int. 2015 Jun;46(6):513-21. doi: 10.3290/j.qi.a33932. PMID 25918755
- [Background] Ghaderi F, Ahmadbeigi M, Vossoughi M, Sardarian A. The efficacy of administrating a sweet-tasting solution for reducing the pain related to dental injections in children: A randomized controlled trial. Int J Paediatr Dent. 2021 Mar;31(2):184-190. doi: 10.1111/ipd.12697. Epub 2020 Aug 25. PMID 32757418
- [Background] Ghadimi S, Estaki Z, Rahbar P, Shamshiri AR. Effect of visual distraction on children's anxiety during dental treatment: a crossover randomized clinical trial. Eur Arch Paediatr Dent. 2018 Aug;19(4):239-244. doi: 10.1007/s40368-018-0352-x. Epub 2018 Jun 12. PMID 29949082
- [Background] Jones CM, Heidmann J, Gerrish AC. Children's ratings of dental injection and treatment pain, and the influence of the time taken to administer the injection. Int J Paediatr Dent. 1995 Jun;5(2):81-5. doi: 10.1111/j.1365-263x.1995.tb00169.x. PMID 7547818
- [Background] Nuvvula S, Alahari S, Kamatham R, Challa RR. Effect of audiovisual distraction with 3D video glasses on dental anxiety of children experiencing administration of local analgesia: a randomised clinical trial. Eur Arch Paediatr Dent. 2015 Feb;16(1):43-50. doi: 10.1007/s40368-014-0145-9. Epub 2014 Sep 26. PMID 25256207
- [Background] Srouji R, Ratnapalan S, Schneeweiss S. Pain in children: assessment and nonpharmacological management. Int J Pediatr. 2010;2010:474838. doi: 10.1155/2010/474838. Epub 2010 Jul 25. PMID 20706640
- [Background] Pepino YM, Mennella JA. Sucrose-induced analgesia is related to sweet preferences in children but not adults. Pain. 2005 Dec 15;119(1-3):210-218. doi: 10.1016/j.pain.2005.09.029. Epub 2005 Nov 18. PMID 16298489